CLINICAL TRIAL: NCT07279194
Title: Efficacy and Safety of HDM1005 Once Weekly in Chinese Participants Without Type 2 Diabetes Who Have Obesity or Are Overweight With Weight-Related Comorbidities: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of HDM1005 in Chinese Obesity or Overweight Patients Without Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM1005-301
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HDM1005 Cohort 1 (Experimental)
  Interventions: Drug: HDM1005 1
- HDM1005 Cohort 2 (Experimental)
  Interventions: Drug: HDM1005 2
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HDM1005 1 — Initiate at a once weekly dose of 0.5 mg and followed a dose escalation regimen, with dose increases every 4 weeks aiming at reaching the maintenance dose, the intervention will last for 52 weeks in total.
  Arms: HDM1005 Cohort 1
Drug: HDM1005 2 — Initiate at a once weekly dose of 0.5 mg and followed a dose escalation regimen, with dose increases every 4 weeks aiming at reaching the maintenance dose. The intervention will last for 52 weeks in total.
  Arms: HDM1005 Cohort 2
Drug: Placebo — Initiate at a once weekly dose of 0.5 mg and followed a dose escalation regimen, with dose increases every 4 weeks aiming at reaching the maintenance dose. The intervention will last for 52 weeks in total.
  Arms: Placebo

SUMMARY:
This is a 56-week randomized, double blinded, parallel-controlled study evaluating the efficacy andsafety of the HDM1005 in patients with obesity or overweight. Eligible participants will be screened and randomized to different dose group of HDM1005 or the placebo group at a ratio of 1:1:1 , HDM1005 or placebo will be given once weekly for 52 weeks, following by a safety follow up of 4 weeks. All participants received a lifestyle intervention that involved counselling on diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years at the time of signing informed consent.
2. BMI≥28 kg/m2 or ≥24 kg/m2 and previously diagnosed with at least one of the following weight related comorbidities: hypertension, dyslipidemia, pre-diabetes, obstructive sleep apnea, fatty liver, weight-bearing joint pain.
3. A self-reported change in body weight no more than 5% within 90 days before screening.
4. Able to understand the procedures and methods of this study, willing to strictly comply with the clinical trial protocol to complete this trial, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Have type 1 diabetes mellitus (T1DM) or T2DM.
2. Have HbA1c≥6.5% or fasting serum glucose (FSG)≥7.0 mmol/L at Visit 1.
3. Have obesity induced by other endocrinologic disorders (for example, Cushing syndrome) or by other medicine.
4. Use of GLP-1 receptor (GLP-1R) agonists or GLP-1R/GCGR agonists or GIPR/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists within 3 months prior to screening.
5. Use of hypoglycemic drugs within 3 months prior to screening.
6. History of thyroid C-cell carcinoma, multiple endocrine neoplasia (MEN) 2A or 2B or relevant family history.
7. Previous history of acute and chronic pancreatitis, acute gallbladder disease history (except cholecystectomy) history.
8. PHQ questionnaire ≥ 15 points at screening or randomization.
9. Have had a history of moderate to severe depression; Or have a history of severe mental illness in the past.
10. Uncontrolled hypertension prior to screening, defined as: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg (stable for 1 month if using antihypertensive drugs).
11. History of malignancy (except cured basal cell carcinoma) in the past 5 years or at the time of screening.
12. History of severe cardiovascular or cerebrovascular diseases within the past six months.
13. History of alcohol and drug abuse at screening.
14. The participant may be allergic to ingredients in the study drug or drugs of the same class.
15. Pregnant or lactating females, males or females of childbearing potential not willing to use contraception throughout the study.
16. The subject has any other factors that may affect the efficacy or safety evaluation of this study, and is not suitable for participation in this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female aged 18 years or above at the time of signing the informed consent
Enrollment: 825 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
primary outcome | week 40
  The percentage change in body weight from baseline to week 40
Co-primary outcome | week 40
  Proportion of subjects with body weight reduction ≥ 5% at Week 40.

SECONDARY OUTCOMES:
secondary outcome | week 40
  The proportion of participants reaching a body weight loss of at least 10% and 15% at week 40
secondary outcome | week 40
  Change in waist circumference, body weight and BMI at week 40
secondary outcome | week 52
  Change in waist circumference, body weight and BMI at week 52
secondary outcome | week 40
  Change in systolic blood pressure (SBP), diastolic blood pressure (DBP) and lipids at week 40
secondary outcome | week 52
  Change in SBP, DBP and lipids at week 52
safety outcome | week 52
  the incidence of adverse events
patient report outcome | week 52
  36-Item Short Form Health Survey, Version 2 questionnaire (scores range from 0 to 100, with higher scores indicating better health status) after administration for 52 weeks.
Immunogenicity outcome | week 52
  ADA and NAb

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hoapital, Shanghai, China